CLINICAL TRIAL: NCT01284673
Title: Characterization of the Cord Blood Stem Cell in Situation of Neonatal Asphyxia
Acronym: NEOCORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-A00076-33
Record Dates: First submitted 2010-04-16; First posted 2011-01-27 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: Cord blood stem; neonatal asphyxia
MeSH Terms: conditions — Respiratory Distress Syndrome; Asphyxia Neonatorum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: in vitro characterization of the cord blood stem cell — The quantitative and qualitative, functional characterization will insist on cell populations which could potentially participate to neuronal regeneration. and assessment such characteristics in conditions of cryo-preservation, compared to fresh cell preparation

SUMMARY:
Neonatal anoxic-ischaemic enkephalopathy is a dramatic perinatal complication due to brain asphyxia. Neurological and neurosensory sequelae are frequent in survivors, due to neuronal damage and loss.

For the moment, only total or partial body hypothermia can partially prevent cell loss. However, no treatment exists to restore neuronal functions.

Cord blood stem cells are a promising treatment for the near future. However, before conducting a clinical trial to evaluate the safety and feasibility of autologous cell therapy in neonatal asphyxia, in vitro characterization of the cord blood stem cell in situation of neonatal asphyxia, compared to normal situation, is needed.

The primary objective of this study is to characterize cord blood stem cells of neonates with neonatal asphyxia and to compare them with those from healthy newborn. The quantitative and qualitative, functional characterization will insist on cell populations which could potentially participate to neuronal regeneration. Secondary objectives are to assess such characteristics in conditions of cryo-preservation, compared to fresh cell preparation

DETAILED DESCRIPTION:
Methods :

Descriptive, bi-centre study on 10 cord blood samples from newborn infants with neonatal asphyxia (5) according to pre-defined criteria, compared healthy neonates (5). The total duration of the study will be 2 years. Parents will be informed and a signed parental consent will be asked in the hours following birth before the in vitro study.

Biological analysis will include elementary analyses for cell quality control, endothelial progenitor exploration, and investigation of mesenchymal stem cells function and of their neuronal differentiation potential (on fresh and frozen samples).

Statistical analysis: comparison between the 2 groups (neonatal asphyxia versus control) would use non parametric test (Mann-Whitney)

This study will allow to evaluate the therapeutic potential of cord blood stem cells autologous transplantation in neonatal asphyxia. It will contribute to the determination of the feasibility of a clinical trail of autologous, cord blood stem cells therapy in such disease.

ELIGIBILITY:
Inclusion Criteria:

* delivery at 37 week or more of pregnancy
* normal pregnancy and delivery

Exclusion Criteria:

* parental refusal

Ages: 1 Minute to 20 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2010-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to characterize cord blood stem cells of neonates with neonatal asphyxia and to compare them with those from healthy newborn | two years
  The quantitative and qualitative, functional characterization will insist on cell populations which could potentially participate to neuronal regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Umberto SIMEONI, MD PhD, Principal Investigator — AP-HM
Locations (1):
- Assistance publique Hopitaux de Marseille, Marseille, bouches du Rhone, France